CLINICAL TRIAL: NCT01443312
Title: Demographic, Clinical, Laboratory and Genetical Characteristics of Patients With Beta Thalassemia Intermedia
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Dpt B and Pediatric Hematology Unit, HaEmek Medical Center, Israel
Other Study IDs: 0047-10-EMC
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Thalassemia
Keywords: Beta globin gene; Alfa globin gene; xmn1 polymorphism
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples will be obtained to analyze the beta and alfa globin genes and the xmn1 polymorphism.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thalassemia Intermedia Patients: Patients with Beta Thalassemia Intermedia treated at the Pediatric Hematology Unit. The characterization of Thalassemia Intermedia was based on age at diagnosis (Older than 2 ys) and / or clinical characteristics that are milder than Thalassemia Major in patients homozygous for beta globin genes.
  Interventions: Genetic: Laboratory analysis.

INTERVENTIONS:
Genetic: Laboratory analysis. — The blood transfusions given to the patients are in accord to physician decision and not related to the study

SUMMARY:
The definition of Thalassemia Intermedia is not generally accepted and the specific clinical and laboratory characteristics varies between patients. Some patients are blood transfusion dependent and others are occasionally transfused. Also the mutations in the beta globin gene are diverse. Another mutations including mutations in the alfa globin gene and in the xmn1 gene can affect the clinical course of this disease. The purpose of this study is to summarize the characteristics of patients with Thalassemia Intermedia treated at the Pediatric Hematology Unit at the HaEmek Medical Center in Israel

DETAILED DESCRIPTION:
The characteristics that will be recorded from the medical files include: demographic data, included gender and ethnic origin, family history, age at diagnosis, number and frequency of blood transfusions including age of first transfusion and physical examination findings.

The laboratory data included iron metabolism parameters, mutation in the alfa and beta gene and the presence of the xmn1 polymorphism.

ELIGIBILITY:
Inclusion Criteria:

-All patients treated at the Pediatric Hematology Unit

Exclusion Criteria:

* Not enough medical records.
* Patients who refuse to give consent to perform genetic studies will be included in the study but only the retrospective clinical data will be recorded.

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with beta Thalassemia Intermedia.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The characteristics of patients with thalassemia intermedia | One year
  Observational study that analyzed the characteristics of thalassemia intermedia patients

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Principal Investigator — Ha'Emek Medical Center, Afula, Israel
Locations (1):
- Pediatric Hematology Unit - Ha'Emek Medical Center, Afula, Israel